CLINICAL TRIAL: NCT01139723
Title: A Phase I, Open Label, Dose Escalation Study of the Safety and Pharmacokinetics of MINT1526A, Administered Intravenously As a Single Agent and in Combination With Bevacizumab to Patients With Advanced Solid Tumors
Brief Title: A Study of the Safety and Pharmacokinetics of MINT1526A, Administered Intravenously As a Single Agent and in Combination With Bevacizumab to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNT4863g; GO00808 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers
MeSH Terms: interventions — Bevacizumab

ARMS (2):
- A (Experimental)
  Interventions: Drug: MINT1526A
- B (Experimental)
  Interventions: Drug: MINT1526A; Drug: bevacizumab

INTERVENTIONS:
Drug: MINT1526A — Intravenous escalating dose
Drug: bevacizumab — Intravenous repeating dose
  Arms: B

SUMMARY:
This is a Phase I, first-in-human, open label, dose-escalation study of MINT1526A administered alone and in combination with bevacizumab by IV infusion every 3 weeks to patients with advanced solid tumors for whom standard therapy either does not exist or has proven to be ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable, or metastatic solid malignancy that has progressed on or failed to respond to regimens or therapies known to provide clinical benefit
* Adequate hematologic and end organ function
* Evaluable disease or measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.0; prostate cancer patients with nonevaluable or nonmeasurable disease if they have an increase in prostate-specific antigen (PSA); ovarian cancer patients with nonevaluable or nonmeasurable disease if they have an increase in cancer antigen 125 (CA-125)
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement to use an effective form of contraception and to continue its use for 6 months after discontinuation from the study

Exclusion Criteria:

* Any anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy within a specified timeframe prior to initiation of study treatment.
* Leptomeningeal disease
* Active infection requiring intravenous antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs, inhaled corticosteroids, or prednisone
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, or cirrhosis
* Known primary central nervous system (CNS) malignancy or untreated or active CNS metastases
* Pregnancy, lactation, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Days 1 to 21 of cycle 1
Incidence, nature, and severity of adverse events and serious adverse events, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v4.0 | Day 1 to study completion

SECONDARY OUTCOMES:
Pharmacokinetic parameters of MINT1526A (including total exposure, maximum and minimum serum concentration, clearance, volume of distribution at steady state) | Following administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Ina Rhee, M.D., Study Director — Genentech, Inc.
Locations (3):
- United States (3):
  - Encinitas, California
  - Los Angeles, California
  - Aurora, Colorado